CLINICAL TRIAL: NCT06179316
Title: The Relationship Between Bone Pelvis Measurements and Erectile Function in Patients Who Had Nerve-Sparing Robot-Assisted Radical Prostatectomy Operation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, principle investigator, Ankara Training and Research Hospital
Other Study IDs: AŞH.AKYILDIZ.007
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- preoperative patients
  Interventions: Procedure: Robot Assisted Radical Prostatectomy
- Patients in the 3rd postoperative month
- Patients in the 6th month postoperatively

INTERVENTIONS:
Procedure: Robot Assisted Radical Prostatectomy — Performing radical prostatectomy operation using robotic equipment while preserving bilateral nerve bundles
  Other Names: Bilateral Nerve-Sparing Robot-Assisted Radical Prostatectomy Operation
  Groups: preoperative patients

SUMMARY:
In order to evaluate the relationship between bone pelvis measurements and erectile function in patients who underwent nerve-sparing robot-assisted radical prostatectomy, bone pelvis measurements will be measured from MRI images of the patients before the operation and their erection quality will be evaluated with the IIEF-5 form. The erection quality of the same patients will be evaluated with the IIEF-5 form in the 3rd and 6th months after the operation. And it will be evaluated whether there is a relationship between the erection quality of the patients before and after the operation and their bone pelvis measurements.

ELIGIBILITY:
Inclusion Criteria:

* Having bilateral nerve-sparing robot-assisted radical prostatectomy operation
* Having a regular sexual life

Exclusion Criteria:

* Having received neoadjuvant therapy
* Having a history of radiotherapy to the pelvic area
* The need to receive postoperative hormono-radiotherapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preoperative Prostate MRI imaging was performed, "Bilateral Nerve Saving Robot Assisted Radical Prostatectomy Operation" was performed, and a regular sexual life was performed; Male patients who have not received neoadjuvant therapy, have no history of radiotherapy to the pelvic region, and do not need postoperative hormono-radiotherapy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
ııef-5 score | three months
  The scale we use to evaluate patients' erection quality